CLINICAL TRIAL: NCT04894916
Title: The My Diabetes Care Patient Portal Intervention for Mobile Devices: A Usability Study
Brief Title: My Diabetes Care Mobile: A Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202268; 1R03DK119735 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Self-efficacy; Patient Web Portals
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Diabetes Care Mobile (MDC-m) (Experimental): Patients have access to a patient web portal embedded with the My Diabetes Care Mobile (MDC-m) intervention.
  Interventions: Other: My Diabetes Care Mobile (MDC-m)

INTERVENTIONS:
Other: My Diabetes Care Mobile (MDC-m) — My Diabetes Care (MDC) is a multi-faceted patient portal intervention for mobile devices that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL), incorporates motivational strategies and access to an online patient support community, and provides literacy level-appropriate and tailored diabetes self-care information.
  Other Names: Patient-facing Diabetes Dashboard

SUMMARY:
The purpose of this study is to conduct a prospective, longitudinal study on the My Diabetes Care mobile (MDC-m) intervention to assess usage patterns, user experience, and to uncover errors in functionality prior to a larger interventional trial.

DETAILED DESCRIPTION:
Up to 65 adult patients with type 2 diabetes mellitus will be enrolled and given access to My Diabetes Care mobile (MDC-m). My Diabetes Care mobile (MDC-m) is a multi-faceted patient portal intervention for mobile devices that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL), incorporates motivational strategies and access to an online patient support community, and provides literacy level-appropriate and tailored diabetes self-care information. Patients will be invited by mail to be screened for enrollment in the study. Interested patients will be able to complete an electronic consent form and enroll online via Research Electronic Data Capture (REDCap™) version 5.0.8. Study participants will complete questionnaires electronically via email using REDCap™ at two time points: baseline (T0) and one-month follow-up (T1). Participants will complete an baseline questionnaire (T0) including basic demographic questions, items about computer usage and internet access, and validated measures of health literacy and eHealth literacy. Each participant will have access to the MDC-m for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Currently taking at least one medication for diabetes
* Age 21 or over
* Able to speak and read in English
* Reliable access to a smartphone or tablet with internet access
* Active VUMC patient web portal (known as My Health At Vanderbilt) account

Exclusion Criteria:

* Residing in a long term care facility
* Medical condition that affects my memory or ability to think.
* Severe visual impairment
* Patients with unintelligible speech (e.g., dysarthria)
* Currently participating in another diabetes-related research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published in a peer-reviewed journal, de-identified individual participant data that underlie the results reported will be available upon requests made to the principal investigator and ending after 36 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data that underlie the results reported will be available after publication in a peer reviewed journal and posted on clinical trials and ending after 36 months after publication.
Access Criteria: Researchers should provide a methodologically sound proposal to achieve their proposed aims. Proposals may be submitted to the principal investigator up to 36 months following publication. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 64 enrolled participants, 59 completed the baseline questionnaire and were with given access to the intervention (My Diabetes Care).
Period: Overall Study
Arm/Group | My Diabetes Care Mobile (MDC-m)
Started | 59
Completed | 53
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32
  Black | 21
  American Indian / Alaska Native | 1
  Asian | 2
  More than one race | 2
  Other | 1
Education [Count of Participants; unit: Participants]
  High school graduate or GED | 5
  Some college or technical school | 14
  College graduate | 16
  Some graduate school/work | 6
  Graduate degree | 18
Employment [Count of Participants; unit: Participants]
  Full time | 23
  Part time | 4
  Unemployed/laid off, looking for work | 1
  Retired | 21
  Disabled, not able to work | 7
  Others | 3
Health Literacy [Count of Participants; unit: Participants] — Health literacy was assessed using a validated one-item screener that asked respondents to rate their confidence independently filling out medical forms on a scale ranging from 'extremely' to 'not at all' confident. Consistent with prior studies, we categorized participants noting any lack of confidence filling out medical forms as having limited health literacy.
  Participants
    Adequate | 51
    Limited | 8
eHealth Literacy [Mean (Standard Deviation); unit: units on a scale] — eHealth refers to healthcare services provided electronically via the Internet. eHealth Literacy refers to the knowledge, comfort, and perceived skill at finding, evaluating, and applying electronic health information to health problems. eHealth Literacy was assessed by the eHEALS scale which contains 8 items, measured with a 5-point Likert scale with response options ranging from "strongly disagree=1" to "strongly agree=5." Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
  units on a scale | 32.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Usability
Description: The System Usability Scale (SUS) is a valid measure of usability and assesses users' perceptions of ease of use, likability of the interface, and overall satisfaction using a 5- point Likert scale (strongly disagree to strongly agree). The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 85 or above suggests excellent usability. The SUS has been used in several studies of patient facing health information technology (the article describing its psychometric properties has been cited over 500 times) and has excellent internal consistency reliability (Cronbach's alpha of 0.91).
Time Frame: One-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the System Usability Scale items on the post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 52
score on a scale | 81.9 (15.4)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); One-sample t-test comparing the sample mean to the threshold value of 71 indicative of "good" usability. The null hypothesis: true mean is equal to 71; Test type: Other — single group; p < 0.001, t-test, 2 sided; mean = 81.9

2. Primary Outcome: System Usage Data
Description: Self-reported usage of My Diabetes Care to include total number of participants who visited MDC-m during the study period and total number of participants with who used MDC-m for 10 minutes or more during the study period.
Time Frame: One-month follow-up
Population: Number analyzed includes only participants that answered the survey items. One participant did not answer the items.
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 58
Participants
  Did you use My Diabetes Care during the study period?: Yes | 54
  Did you use My Diabetes Care during the study period?: No | 4
  Did you use My Diabetes Care for 10 minutes or more?: Yes | 47
  Did you use My Diabetes Care for 10 minutes or more?: No | 11

3. Primary Outcome: User Experience
Description: Unique study specific items to assess participants' perspectives on the usefulness of particular My Diabetes Care features and functionality.
Time Frame: One-month follow-up
Measure: Number; unit: participants
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 53
participants
  Question Mark Icon - useful | 25
  Goal, Caution, and Warning Ranges - useful | 40
  Graphs showing trends in your diabetes health data over time - useful | 41
  Patients Like Me Data - useful | 25
  Literacy level appropriate educational links about each diabetes health measure - useful | 24
  Make a Change for the Better module - useful | 21
  Literacy level appropriate educational links with tips to improve your diabetes - useful | 22
  Diabetes Online Community - useful | 8

4. Secondary Outcome: Change in Diabetes Knowledge
Description: The Short Diabetes Knowledge Instrument (SDKI) is a valid measure of diabetes knowledge with an emphasis on controlling blood glucose through diet, recognizing symptoms of abnormal blood glucose, and using healthy eating to prevent complications. It also includes items on foot care and the importance of physical activity for preventing cardiovascular complications. The SDKI is a uni-dimensional, 13-item scale with scores ranging from 0 to 13 (number of items answered correctly). SDKI demonstrated good internal consistency reliability (Cronbach's alpha 0.73) in a multi-ethnic sample of older adults suggesting the instrument can be used to measure diabetes knowledge in diverse populations (Quandt et al. Diabetes Educator, 2014).
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the Short Diabetes Knowledge Instrument items on the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 49
score on a scale
  Baseline pre-questionnaire | 5.37 (1.6)
  One-month follow-up post-questionnaire | 6.10 (1.5)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 0.73

5. Secondary Outcome: Change in Diabetes Self-Efficacy
Description: The Perceived Diabetes Self-Management Scale (PDSMS) is a valid measure of diabetes self-efficacy (i.e., how confident they feel about their ability to carry out multiple self management tasks). The uni-dimensional, 8-item scale is scored on a five-point Likert scale. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the Perceived Diabetes Self-Management Scale items on the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 50
score on a scale
  Baseline pre-questionnaire | 29.12 (5.1)
  One-month follow-up post-questionnaire | 30.29 (5.2)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.08, t-test, 2 sided; Mean Difference (Net) = 1.17

6. Secondary Outcome: Change in Number of Participants That Correctly Identified Definitions and Goal Ranges for Diabetes Health Measures
Description: Unique study specific items to assess participants' knowledge of measures of diabetes health status (i.e., Hemoglobin A1C, blood pressure, low-density lipoprotein, and flu vaccination status). Each multiple choice item has one correct answer and the unit of measure is the number of participants that correctly answered each item.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the Knowledge of Diabetes Measures items on the pre- and post-questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 53
Participants
  Identify definition of A1c at baseline | 49
  Identify definition of A1c at one-month follow-up | 51
  Identify goal range for A1c at baseline | 30
  Identify goal range for A1c at one-month follow-up | 36
  Identify definition of blood pressure at baseline | 36
  Identify definition of blood pressure at one-month follow-up | 41
  Identify goal range for blood pressure at baseline | 16
  Identify goal range for blood pressure at one-month follow-up | 23
  Identify definition of LDL cholesterol at baseline | 32
  Identify definition of LDL cholesterol at one-month follow-up | 38
  Identify goal range for LDL cholesterol at baseline | 22
  Identify goal range for LDL cholesterol at one-month follow-up | 27
  Identify definition of flu vaccine at baseline | 52
  Identify definition of flu vaccine at one-month follow-up | 53
  Identify frequency of flu vaccination at baseline | 48
  Identify frequency of flu vaccination at one-month follow-up | 51
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Analysis for pre-post change in knowledge of definition of A1C; Test type: Other; p = 0.68, McNemar
Statistical Analysis 2: Comparison: My Diabetes Care Mobile (MDC-m); Analysis for pre-post change in knowledge of goal range for hemoglobin A1c; Test type: Other; p = 0.18, McNemar
Statistical Analysis 3: Comparison: My Diabetes Care Mobile (MDC-m); Analysis for pre-post change in knowledge of definition of systolic blood pressure; Test type: Other; p = 0.18, McNemar
Statistical Analysis 4: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in knowledge of goal range for systolic blood pressure; Test type: Other; p = 0.17, McNemar
Statistical Analysis 5: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in knowledge of definition of LDL cholesterol; Test type: Other; p = 0.33, McNemar
Statistical Analysis 6: Comparison: My Diabetes Care Mobile (MDC-m); Analysis for pre-post change in knowledge of goal range for LDL cholesterol; Test type: Other; p = 0.40, McNemar
Statistical Analysis 7: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in knowledge of definition of flu vaccine; Test type: Other; p = 1.00, McNemar
Statistical Analysis 8: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in knowledge of recommended frequency of flu vaccination; Test type: Other; p = 0.37, McNemar

7. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. The five-item, uni-dimensional scale has scores that range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress. The PAID-5 has excellent excellent internal consistency reliability (Cronbach's alpha 0.86) and is associated with measures of depression and hemoglobin A1c.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the Problem Areas in Diabetes Scale (PAID-5) items on the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 50
score on a scale
  Baseline pre-questionnaire | 4.92 (4.7)
  One-month follow-up post-questionnaire | 4.21 (3.8)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.16, t-test, 2 sided; Mean Difference (Net) = -0.71

8. Secondary Outcome: Change in Diabetes Attitudes
Description: Unique study specific items to assess participants' attitudes toward social comparisons (2 items) and goal-based comparisons (2 items) regarding their diabetes health status. Each items is scored on a 5-point Likert scale from '1=strongly disagree' to '5=strongly agree'.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered the study specific diabetes attitudes item on both the pre- and post-questionnaire.
Measure: Number; unit: participants
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 53
participants
  Interested in social comparison info at baseline - Strongly Agree/Agree | 43
  Interested in social comparison info at one-month follow-up -Strongly Agree/Agree | 33
  Interested goal-based comparison info at baseline -Strongly Agree/Agree | 50
  Interested goal-based comparison info at one-month follow-up -Strongly Agree/Agree | 47
  Social comparison info is useful at baseline - Strongly Agree/Agree | 50
  Social comparison info is useful at one-month - Strongly Agree/Agree | 47
  Goal-based comparison info is useful at baseline - Strongly Agree/Agree | 51
  Goal-based comparison info is useful at one-month - Strongly Agree/Agree | 49
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in interest in information about how my diabetes health data compares to other patients like me (i.e., social comparison information); Test type: Other; p = 0.03, McNemar
Statistical Analysis 2: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in interest in information about how their diabetes health data compares to the goal range (i.e., goal-based comparison information); Test type: Other; p = 0.45, McNemar
Statistical Analysis 3: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in agreement with statement: 'Information about how my diabetes health data compares to other patients like me [social comparison information] is useful; Test type: Other; p = 0.17, McNemar
Statistical Analysis 4: Comparison: My Diabetes Care Mobile (MDC-m); Analysis of pre-post change in agreement with statement: 'Information about how my diabetes health data compares to the goals range [goal-based comparison information] is useful; Test type: Other; p = 0.62, McNemar

9. Secondary Outcome: Change in Diabetes Readiness for Change
Description: Four-item assessment of stage of change based on the Transtheoretical Model (TTM) of behavior change. It includes questions one item each assessing the participants stage of change for: (1) physical activity, (2) medication management, (3) glucose self-monitoring, and (4) diet. There are five response options per item that categorize the participants' current TTM stage of change for the item: (a) Precontemplation, (b) Contemplation, (c) Preparation, (d) Action, and (e) Maintenance.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires)
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 53
Participants
  Pre-intervention: Taking Medicines: Precontemplation | 0
  Pre-intervention: Taking Medicines: Contemplation | 0
  Pre-intervention: Taking Medicines: Preparation | 1
  Pre-intervention: Taking Medicines: Action | 6
  Pre-intervention: Taking Medicines: Maintenance | 46
  Pre-intervention: Taking Medicines: Missing/No Answer | 0
  Post-intervention: Taking Medications: Precontemplation | 1
  Post-intervention: Taking Medications: Contemplation | 0
  Post-intervention: Taking Medications: Preparation | 1
  Post-intervention: Taking Medications: Action | 3
  Post-intervention: Taking Medications: Maintenance | 48
  Post-intervention: Taking Medications: Missing/No Answer | 0
  Pre-intervention: Exercising: Precontemplation | 9
  Pre-intervention: Exercising: Contemplation | 10
  Pre-intervention: Exercising: Preparation | 9
  Pre-intervention: Exercising: Action | 11
  Pre-intervention: Exercising: Maintenance | 14
  Pre-intervention: Exercising: Missing/No Answer | 0
  Post-intervention: Exercising: Precontemplation | 10
  Post-intervention: Exercising: Contemplation | 8
  Post-intervention: Exercising: Preparation | 5
  Post-intervention: Exercising: Action | 14
  Post-intervention: Exercising: Maintenance | 16
  Post-intervention: Exercising: Missing/No Answer | 0
  Pre-intervention: Eating Healthy: Precontemplation | 4
  Pre-intervention: Eating Healthy: Contemplation | 7
  Pre-intervention: Eating Healthy: Preparation | 9
  Pre-intervention: Eating Healthy: Action | 12
  Pre-intervention: Eating Healthy: Maintenance | 21
  Pre-intervention: Eating Healthy: Missing/No Answer | 0
  Post-intervention: Healthy Eating: Precontemplation | 7
  Post-intervention: Healthy Eating: Contemplation | 7
  Post-intervention: Healthy Eating: Preparation | 5
  Post-intervention: Healthy Eating: Action | 9
  Post-intervention: Healthy Eating: Maintenance | 24
  Post-intervention: Healthy Eating: Missing/No Answer | 1
  Pre-intervention: Home Glucose Monitoring: Precontemplation | 7
  Pre-intervention: Home Glucose Monitoring: Contemplation | 3
  Pre-intervention: Home Glucose Monitoring: Preparation | 4
  Pre-intervention: Home Glucose Monitoring: Action | 11
  Pre-intervention: Home Glucose Monitoring: Maintenance | 28
  Pre-intervention: Home Glucose Monitoring: Missing/No Answer | 0
  Post-intervention: Home Glucose Monitoring: Precontemplation | 8
  Post-intervention: Home Glucose Monitoring: Contemplation | 2
  Post-intervention: Home Glucose Monitoring: Preparation | 1
  Post-intervention: Home Glucose Monitoring: Action | 11
  Post-intervention: Home Glucose Monitoring: Maintenance | 31
  Post-intervention: Home Glucose Monitoring: Missing/No Answer | 0

10. Secondary Outcome: Change in Diabetes Self-Care (General Diet Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The general diet subscale is used to assess general diet adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "How many of the last SEVEN DAYS have you followed a healthful eating plan?" The general diet subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the items on the Summary of Diabetes Self-Care Activity - General Diet Subscale on both the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 51
score on a scale
  Baseline pre-questionnaire | 4.74 (1.6)
  One-month follow-up post-questionnaire | 4.83 (1.6)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.53, t-test, 2 sided; Mean Difference (Net) = 0.09

11. Secondary Outcome: Change in Diabetes Self-Care (Specific Diet Adherence)
Description: as for outcome 10
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the items on the Summary of Diabetes Self-Care Activity - Specific Diet Subscale on both the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 51
score on a scale
  Baseline Pre-Questionnaire | 4.30 (1.6)
  One-month Follow-up Post-Questionnaire | 4.33 (1.6)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.86, t-test, 2 sided; Mean Difference (Net) = 0.03

12. Secondary Outcome: Change in Diabetes Self-Care (Exercise Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The exercise subscale is used to assess exercise adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "On how many of the last SEVEN DAYS did you participate in at least 30 minutes of physical activity?" The exercise subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the items on the Summary of Diabetes Self-Care Activity - Exercise Subscale on both the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 51
score on a scale
  Baseline Pre-Questionnaire | 3.17 (2.1)
  One-month Follow-up Post-Questionnaire | 3.45 (2.2)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.22, t-test, 2 sided; Mean Difference (Net) = 0.28

13. Secondary Outcome: Change in Diabetes Self-Care (Self-Monitoring of Blood Glucose Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The blood-glucose testing subscale is used to assess self-monitoring of blood glucose adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "On how many of the last SEVEN DAYS did you test your blood sugar?" The blood-glucose testing subscale is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline to one-month Follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the items on the Summary of Diabetes Self-Care Activity - Blood-glucose Testing Subscale on both the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 51
score on a scale
  Baseline Pre-Questionnaire | 4.05 (2.9)
  One-month Follow-up Post-Questionnaire | 4.3 (2.7)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.21, t-test, 2 sided; Mean Difference (Net) = 0.25

14. Secondary Outcome: Change in Medication Adherence
Description: The Adherence to Refills and Medications Scale is a reliable and valid measure of medication adherence. The 12-item ARMS has good internal consistency reliability (α=0.81). Responses range from 1="none of the time" to 4="all of the time," and are summed to produce an overall adherence score ranging from 12-48, with higher scores representing more problems with medication adherence.
Time Frame: Baseline to one-month follow-up
Population: Participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires) AND answered all the Adherence to Refills and Medications Scale items on the pre- and post-questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | My Diabetes Care Mobile (MDC-m)
Number analyzed (Participants) | 47
score on a scale
  Baseline pre-questionnaire | 14.12 (3.5)
  One-month follow-up post-questionnaire | 13.73 (3.3)
Statistical Analysis 1: Comparison: My Diabetes Care Mobile (MDC-m); Test type: Other; p = 0.18, t-test, 2 sided; Mean Difference (Net) = -0.39

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | My Diabetes Care Mobile (MDC-m)
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04894916/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04894916/ICF_000.pdf